CLINICAL TRIAL: NCT00168714
Title: Avonex Pregnancy Exposure Registry
Brief Title: Pregnancy Exposure Registry for Avonex (Interferon Beta-1a)
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: C-871
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Prenatal Exposure Delayed Effects; Multiple Sclerosis; Pregnancy
Keywords: AVONEX; Pregnancy
MeSH Terms: conditions — Prenatal Exposure Delayed Effects; Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pregnant participants: Pregnant participants who were exposed to Avonex within approximately 1 week of conception or during the first trimester of pregnancy
  Interventions: Drug: BG9418 (interferon beta-1a)

INTERVENTIONS:
Drug: BG9418 (interferon beta-1a) — Exposure to Avonex during pregnancy
  Other Names: Avonex

SUMMARY:
The primary objectives of the study were to prospectively record and analyze birth defects and spontaneous fetal losses in women with multiple sclerosis (MS) exposed to Avonex within approximately 1 week of conception or during the first trimester of pregnancy, where the outcome of the pregnancy was unknown prospectively and to prospectively record and analyze pregnancy outcomes in an exploratory fashion of women with MS who stopped therapy, but who may have been exposed to Avonex with approximately 1 week of conception or during the first trimester of pregnancy.

ELIGIBILITY:
Key Inclusion Criteria:

* Have been exposed to AVONEX within approximately 1 week of conception or during the first trimester of pregnancy.
* Provide sufficient information to determine that the pregnancy is prospectively registered (i.e., the outcome of pregnancy must be unknown prospectively).
* Provide verbal consent to participate in the Registry.
* Verbally provide contact information for herself, her HCP, and the infant's HCP (if applicable).

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with MS who were exposed to Avonex in the US
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2004-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Record and analyze birth defects and spontaneous fetal losses | Prospectively, MS women exposed to Avonex within 1 week of conception or during the first trimester of pregnancy
Record and analyze pregnancy outcomes | Prospectively, MS women who stopped therapy, but may have been exposed to Avonex within 1 week of conception or during the first trimester of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Kendle, Wilmington, North Carolina, United States

REFERENCES:
- [Derived] Weinstock-Guttman B, Ross AP, Planton J, White K, Pandhi A, Greco A, Kumar A, Everage N, Vignos M. Analysis of Pregnancy Outcomes Following Exposure to Intramuscular Interferon Beta-1a: The AVONEX(R) Pregnancy Exposure Registry. Drugs Real World Outcomes. 2023 Dec;10(4):503-511. doi: 10.1007/s40801-023-00384-0. Epub 2023 Sep 22. PMID 37737962